CLINICAL TRIAL: NCT05750810
Title: Exacerbations and Their Outcomes International (EXACOS International): Burden of Severe Exacerbations of COPD and the Association Between Frequency of Severe Exacerbations and Clinical and Health-care Utilization Outcomes
Brief Title: Exacerbations and Their Outcomes International (EXACOS International)
Status: Completed | Type: Observational
Sponsor: Joon Young Choi (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Hallym University Medical Center (Other); Konkuk University Hospital (Other)
Responsible Party: Sponsor-Investigator, Joon Young Choi, Clinical assistant professor, Incheon St.Mary's Hospital
Organization: Incheon St.Mary's Hospital (Other)
Other Study IDs: ESR-21-21659
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: COPD; Exacerbation Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Severe exacerbation frequency — A severe exacerbation will be primarily defined as a hospitalization (with or without ICU) or an emergency department visit as a result of worsening of COPD symptoms.

SUMMARY:
The aim of this study is to quantify the burden of severe AECOPD in South Korea, by investigating the association between frequency of severe AECOPD and clinical and health-care utilization outcomes.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE Chronic obstructive pulmonary disease (COPD) is a common, progressive disease characterized by airflow obstruction which is not fully reversible. Acute exacerbations of COPD (AECOPD) are worsening of COPD symptoms (breathlessness, cough, and sputum volume and purulence) beyond normal day to day variation. Between 30-50% of patients with COPD experience at least one AECOPD per year [1]. Even a single moderate AECOPD increases risk of future multiple AECOPD events, starting a spiral of excessive disease progression and leading to an increased risk of death [2]. AECOPDs have also been associated with other clinical outcomes such as accelerated lung function decline [3,4].

   Studies have shown that AECOPDs are related to future AECOPDs, however, little is known about clinical burden and health care utilization in the COPD population [2, 5]. To date, most of published literature reports a combined category of moderate-severe exacerbations, typically stratifying patients as experiencing frequent (i.e. two or more events per patient-year) vs. infrequent (none or one) exacerbations.

   The aim of this study is to quantify the burden of severe AECOPD in South Korea, by investigating the association between frequency of severe AECOPD and clinical and health-care utilization outcomes.

   This study will help to understand the relationship between severe AECOPD and clinical and health care utilization burden in South Korea with no established health care databases.
2. OBJECTIVES AND HYPOTHESES The objective is to quantify the burden of severe AECOPD by describing the clinical and health care utilization burden of AECOPD by frequency.

2.1 Primary Objectives

2.1 Primary Objectives & Hypothesises

1. To estimate the frequency of severe AECOPD, in a COPD population
2. To describe any time trends in the frequency of severe exacerbations throughout the study period (over a 2-year period)
3. To describe lung function decline over time (FEV1)
4. To quantify health care resource utilization by number of severe AECOPD over a 2-year period

2.2 Secondary Objective & Hypothesis

1. Modified Medical Research Council (mMRC) dyspnea scale measured at time of the visit

   3. METHODOLOGY

   3.1 Study Design - General Aspects This study was based on the Korea COPD Subgroup Study (KOCOSS) database, constructed from a nationwide prospective cohort study-initiated in April 2012-that involved 54 medical centers in South Korea.

   During the patient visit, data was captured through the use of Case Report Forms (CRFs) by a doctor or trained nurse. After a baseline evaluation, patients were examined at 1-year follow-up.

   3.2 Study Population

   Inclusion criteria of the KOCOSS database is as follows:

   1) Age > 40 years; 2) those with post-bronchodilator (FEV1)/forced vital capacity (FVC) ≤ 70% of the normal predicted value.

   The following subpopulations of interest will be identified:

   • Patients with eosinophils ≥100cells/ul

   • Patients with a history of a comorbidity of special interest:

   - Any history of major cardiovascular comorbidity as recorded in the medical records: AMI, heart failure, stroke (+ MACE)

   - Any cardiovascular risk factor as recorded in the medical history: hypertension, diabetes - Any history of other major comorbidity: depression, anxiety, GERD, renal failure, etc.

   3.3 Study Period Data of COPD patients from April 2012 to 2021 will be extracted and analyzed

   4. VARIABLES AND EPIDEMIOLOGICAL MEASUREMENTS

   4.1 Exposures

   The main exposure for this study is severe exacerbation frequency. A severe exacerbation will be primarily defined as a hospitalization (with or without ICU) or an emergency department visit as a result of worsening of COPD symptoms. The number of severe AECOPD was counted at the initial visit in recall of previous 1-year events, and prospectively measured at 1-year follow up visit. The annual severe AECOPD frequency will be estimated in the 2 years (pre- and post- 1-year of initial visit), and divided by 2. This will guide the categorization of the severe AECOPD frequency. We expect the following categories:

   - 0 events

   - 1 severe event
   * 2 severe events
   * 3 severe events
   * >3 severe events

   The distribution of exacerbations across the entire 2 year period will also be described. In order to fully describe severe AECOPDs and their impact in disease progression, clinical burden, and healthcare costs the following outcomes will be measured:

   1) Clinical burden defined as change in lung function (FEV1) over time 2) Co-morbidities 3) Health care utilization burden will be defined accounting for:

   -number of emergency department visits

   -number of hospitalizations

   -number of ICU episodes

   5. STATISTICAL ANALYSIS PLAN

   5.1 Statistical Methods - General Aspects Summary statistics will be provided for the COPD population overall and by sub-populations noted above. Continuous measures will be described using means and standard deviations and categorical measures will be reported using numbers and proportions. Count variables will be expressed as rates per person-year. Groups will be compared using standard univariate statistical methods, including the chi-square test or the Fisher exact test for categorical variables and the analysis of variance test for continuous variables.

   5.2 Sample Size and Power Calculations No power calculations were performed as the objectives of this study are mostly descriptive in nature.

ELIGIBILITY:
* Inclusion Criteria:

  1. Over 40 years old South Korean COPD patients(Bronchodilator test results FEV1/FVC <0.7)
  2. COPD patients who complain of cough, sputum, dyspnea
  3. Unrelated smoking history
* Exclusion Criteria:

  1. other disease like asthma patients which is similar to COPD symptoms.
  2. patients who is not suitable for pulmonary function test and communication
  3. myocardial infarction or cerebrovascular event within the previous 3 months
  4. pregnants
  5. patients who disagree with registration
  6. rheumatoid patients
  7. cancer patients(including metastatic cancer, leukemia, lymphoma)
  8. irritable bowel syndrome
  9. patients who use systemic steroids over 8 weeks due to other diseases except COPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was based on the Korea COPD Subgroup Study (KOCOSS) database, constructed from a nationwide prospective cohort study-initiated in April 2012-that involved 54 medical centers in South Korea. It was designed to evaluate characteristics of COPD patients in South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 3477 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
the frequency of severe AECOPD | 10-year
  To estimate the frequency of severe AECOPD, in a COPD population
time trends in the frequency of severe exacerbations | 2-year
  To describe any time trends in the frequency of severe exacerbations throughout the study period (over a 2-year period)
lung function decline over time | 3-year
  To describe lung function decline over time (FEV1)
health care resource utilization | 2-year
  To quantify health care resource utilization by number of severe AECOPD over a 2-year period

CONTACTS AND LOCATIONS:
Locations (1):
- Incheon St. Mary's Hospital, Incheon, Gyeongki, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD is not available due to restriction

REFERENCES:
- [Derived] Rhee CK, Choi JY, Park YB, Yoo KH. Clinical Characteristics and Frequency of Chronic Obstructive Pulmonary Disease Exacerbations in Korean Patients: Findings From the KOCOSS Cohort 2012-2021. J Korean Med Sci. 2024 May 20;39(19):e164. doi: 10.3346/jkms.2024.39.e164. PMID 38769923